CLINICAL TRIAL: NCT05518669
Title: Mobile Cone-Beam CT in Combination With Electromagnetic Navigation Bronchoscopy for the Diagnosis of Peripheral Pulmonary Nodules
Brief Title: mCBCT in Combination With ENB for the Diagnosis of PPNs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Other Study IDs: SHCHE202207
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Pulmonary Nodules; Lung Cancer
Keywords: Peripheral Pulmonary Nodules; Diagnosis; Mobile Cone-Beam CT; Electromagnetic Navigation Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral Pulmonary Nodules: Patients with peripheral pulmonary nodules on chest computed tomography suspicion of malignancy who are scheduled to reach the target lesion for diagnosis by mobile cone-beam CT combined with electromagnetic navigation bronchoscopy.
  Interventions: Device: Electromagnetic Navigation Bronchoscopy (superDimension™ Navigation System) and Mobile Cone-Beam CT (Cios Spin)

INTERVENTIONS:
Device: Electromagnetic Navigation Bronchoscopy (superDimension™ Navigation System) and Mobile Cone-Beam CT (Cios Spin) — Subjects with biopsy of peripheral pulmonary nodule using electromagnetic navigation bronchoscopy and mobile cone-beam CT.

SUMMARY:
This study aims to evaluate the clinical value of mobile cone-beam CT (mCBCT) in combination with electromagnetic navigation bronchoscopy for the diagnosis of peripheral pulmonary nodules, and to explore the value of mCBCT in improving the diagnostic yield by calculating the improvement in diagnostic yield of patients before and after mCBCT adjustments.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center observational clinical trial to evaluate the diagnostic value of mobile cone-beam CT (mCBCT) in combination with electromagnetic navigation bronchoscopy for the diagnosis of peripheral pulmonary nodules. The investigators will adjust the position of electromagnetic navigation bronchoscopy base on the intraoperative 3D imaging findings of mCBCT. The value of mCBCT in improving diagnostic yield is explored by comparing the diagnostic yield Post-mCBCT with that of Pre-mCBCT. The Pre-mCBCT diagnostic yield is the proportion of patients diagnosed by electromagnetic navigation bronchoscopy and with no need for adjustment after mCBCT spin confirmed "tool-in-lesion" during the procedure in all enrolled subjects. The Post-mCBCT diagnostic yield is the proportion of diagnosed patients with and without adjustment after mCBCT spin during the procedure in all enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age of 18 years and older
* Chest CT imaging shows the presence of peripheral pulmonary nodules (defined as those lesions that are surrounded by pulmonary parenchyma and located below the segmental bronchus) suspicion of malignancy that need to be confirmed by pathology
* Pulmonary nodules of > 8mm and ≤30 mm in largest dimension
* Patients without contraindications of bronchoscopy
* Patients have good medical adherence and signed informed consent

Exclusion Criteria:

* Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy
* Presence of concomitant endobronchial lesion during the bronchoscopy procedure
* Pre-operative mCBCT spin scan showed no visible lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the presence of pulmonary peripheral nodules on chest CT imaging suspicion of malignancy that need to obtain pathologic diagnosis by transbronchial lung biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield improvement ratio | Up to at least 6 months
  Diagnostic yield improvement ratio, defined as Post-mCBCT diagnostic yield minus Pre-mCBCT diagnostic yield.
  The Pre-mCBCT diagnostic yield, defined as the proportion of patients diagnosed by electromagnetic navigation bronchoscopy and without any adjustment after first time mCBCT spin during the procedure in all enrolled subjects.
  The Post-mCBCT diagnostic yield, defined as the proportion of diagnosed patients including those with and without adjustment after mCBCT spin in all enrolled subjects.
  Diagnostic yield was defined as all instances in which the results of bronchoscopy matched the final diagnoses.

SECONDARY OUTCOMES:
Pre-mCBCT navigational yield | Intra-procedure
  The proportion of patients who was confirmed tool-in-lesion by the first time mCBCT spin and no need for further adjustment in all enrolled subjects.
Post-mCBCT navigational yield | Intra-procedure
  The proportion of patients who was confirmed tool-in-lesion with and without adjustment by mCBCT in all enrolled subjects.
Total radiation dose | Intra-procedure
  Radiation dose from procedure, measured by the dose area product (DAP), defined as the product of dose and beam area (Gy cm^2).
Fluoroscopy time | Intra-procedure
  The fluoroscopy time during the procedure.
Adjustment time | Intra-procedure
  The adjustment time during the procedure, defined as the time between the first mCBCT spin scanning to final spin scanning.
Total operation time | Intra-procedure
  The total operation time was defined as the time from bronchoscope insertion to withdrawal of the glottis.
Factors affecting diagnostic yield | Up to at least 6 months
  The factors affecting diagnostic yield includes the nodule nature, nodule size, nodule location, bronchus sign on CT, etc.
Complication rate | Up to 1 month
  The complications refer to the proportion of serious adverse events related to the procedure during or within 1 month after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casal RF, Sarkiss M, Jones AK, Stewart J, Tam A, Grosu HB, Ost DE, Jimenez CA, Eapen GA. Cone beam computed tomography-guided thin/ultrathin bronchoscopy for diagnosis of peripheral lung nodules: a prospective pilot study. J Thorac Dis. 2018 Dec;10(12):6950-6959. doi: 10.21037/jtd.2018.11.21. PMID 30746241
- [Background] Reisenauer J, Duke JD, Kern R, Fernandez-Bussy S, Edell E. Combining Shape-Sensing Robotic Bronchoscopy With Mobile Three-Dimensional Imaging to Verify Tool-in-Lesion and Overcome Divergence: A Pilot Study. Mayo Clin Proc Innov Qual Outcomes. 2022 Apr 23;6(3):177-185. doi: 10.1016/j.mayocpiqo.2022.02.004. eCollection 2022 Jun. PMID 35509435
- [Background] Hsieh MJ, Chou PL, Fang HY, Wen CT, Chao YK. Single-step localization and excision of small pulmonary nodules using a mobile 3D C-arm. Interact Cardiovasc Thorac Surg. 2021 Nov 22;33(6):885-891. doi: 10.1093/icvts/ivab182. PMID 34291295
- [Background] Chen J, Xie F, Zheng X, Li Y, Liu S, Ma KC, Goto T, Muller T, Chan ED, Sun J. Mobile 3-dimensional (3D) C-arm system-assisted transbronchial biopsy and ablation for ground-glass opacity pulmonary nodules: a case report. Transl Lung Cancer Res. 2021 Jul;10(7):3312-3319. doi: 10.21037/tlcr-21-561. PMID 34430367